CLINICAL TRIAL: NCT06306794
Title: The Effect of Crochet Octopus Use on Pain and Comfort in Endotracheal Aspiration of the Premature Infants
Brief Title: Reducing Pain Levels and Increasing Comfort of Premature Infants During Aspiration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nurgül Tekin (Other)
Responsible Party: Sponsor-Investigator, Nurgül Tekin, Msc, Uludag University
Organization: Uludag University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2011-KAEK-25 2023/12-26
Record Dates: First submitted 2024-02-06; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Pain; Premature Baby 26 to 32 Weeks; Premature Baby 33 to 36 Weeks; Aspiration
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: In the calculation of the sample size, the power level is 80% and the significance level is 5%. It was determined by the statistical expert that the number of babies that should be included for each group is 26 and the total number of babies required for the whole study is 52 when the effect size is determined as 0.8 for the investigation of the difference between the experimental and control groups in terms of the premature infant pain profile (PIPP) variable. Based on aforementioned information, the study sample was determined as 80 preterm infants in which 40 for experimental groups and 40 for control groups. Block randomization method will be applied for the randomization of the groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): During the endotracheal aspiration procedure, the octopus will be given to experimental group 10 minutes before the procedure. Babies will be allowed to touch the octopus for 10 minutes during and after the procedure. Physiologic parameters of the infants before, during and after the procedure will be reported and recorded by camera. According to the video recordings, PIPP-R and PICS scale evaluations of the infants will be made by two research nurses other than the main researcher conducting the study.
  Interventions: Other: crochet octopus
- control group (No Intervention): The routine aspiration application steps of the unit will be applied to the control group without any intervention. Physiologic parameters of the infants before, during and after the procedure will be reported and recorded by camera. According to the video recordings, PIPP-R and PICS scale evaluations of the infants will be made by two research nurses other than the main researcher conducting the study.

INTERVENTIONS:
Other: crochet octopus — During the endotracheal aspiration procedure, the octopus will be given to experimental group 10 minutes before the procedure.
  Arms: experimental group

SUMMARY:
The aim of this study was to investigate the effect of using amigurumi octopus on the pain and comfort of the newborn in premature infants undergoing endotracheal aspiration.

It is a randomized controlled quasi-experimental design. The study will be conducted in the neonatal intensive care unit of Health Sciences University Bursa High Specialization Training and Research Hospital. The population of the study will consist of preterm hospitalized in the neonatal intensive care unit during the period of the conducted study. In the calculation of the sample size, the power level is 80% and the significance level is 5%. It was determined by the statistical expert that the number of babies that should be included for each group is 26 and the total number of babies required for the whole study is 52 when the effect size is determined as 0.8 for the investigation of the difference between the experimental and control groups in terms of the premature infant pain profile (PIPP) variable. Based on aforementioned information, the study sample was determined as 80 preterm infants in which 40 for experimental groups and 40 for control groups. Block randomization method will be applied for the randomization of the groups.

PIPP=Premature Infant Pain Scale and Premature Infant Comfort Scale (PBIQ) will be used as a case report form for the collection of the study data. All the patients included in the study will be intervened by the nurse having a neonatal nursing experience by paying attention to aseptic conditions in accordance with the routine aspiration criteria of the unit. Standardization will be ensured by intervening in all patients with the same application by the same nurse.

During the endotracheal aspiration procedure, the octopus will be given to experimental group 10 minutes before the procedure. Babies will be allowed to touch the octopus for 10 minutes during and after the procedure. Physiologic parameters of the infants before, during and after the procedure will be reported and recorded by camera. According to the video recordings, PIPP-R and PICS scale evaluations of the infants will be made by two research nurses other than the main researcher conducting the study. The routine aspiration application steps of the unit will be applied to the control group without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age range of 26-36 weeks
* The baby should be between postnatal day 0 and 5 (Postnatal day of baby should be between 0 and 5 days.)
* Need for invasive mechanical ventilator support
* Need for endotracheal aspiration
* No analgesic, opioid and sedative medication was applied within the 4 hours before the endotracheal aspiration
* At least 2 hours passed since the last painful procedure

Exclusion Criteria:

* Receiving analgesic medication
* Major congenital anomaly
* Having a pneumothorax tube
* Stage III and intraparenchymal hemorrhage
* Receiving a sedative medication

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
pain in the during endotracheal aspiration | 5 minutes
  To decrease the Premature Infant Pain Scale-Revise score of the experimental group compared to the control group.
  Items in the PIPP-R scale include three behavioral (frowning, squinting eyes, prominence of the nasolobial groove), two physiological (heart rate and oxygen saturation) and two contextual (behavioral status and gestational age) items.
  According to the scale, the highest score is 21 for premature babies and 18 for term newborns. According to the scale scoring, scoring between 0 and 6 indicates that the premature baby has mild pain, between 7 and 12 points indicates that the premature baby has moderate pain, and between 13 and 21 points indicates that the premature baby has severe pain.

SECONDARY OUTCOMES:
comfort in the during endotracheal aspiration | 5 minutes
  To decrease The Premature Infant Comfort Scale score of the experimental group compared to the control group.
  It is a multidimensional scale used to evaluate behavioral and psychological comfort and pain. PBCQ evaluates 7 parameters such as Alertness, Calm/Agitation, Respiratory Status (only in mechanical ventilation support) or Crying (not evaluated because it is scored only in children with spontaneous breathing), Physical Movement, Muscle Tone, Facial Movements and Average Heart Rate. Each item is a 5-point Likert type, scored from 1 to 5, from worst to best.
  According to the scale, 35 indicates the lowest and 7 indicates the highest comfort score. A high score from the scale indicates that the comfort level is low. If the total score obtained is ≥17, it is the cut-off value of the scale, it is the limit value for the baby's comfort level and indicates the need for a pain-reducing intervention.

IPD SHARING:
Plan to Share IPD: No